CLINICAL TRIAL: NCT04917770
Title: The Efficacy and Safety of Sintilimab in Combination With Multimodal Radiotherapy in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma After Multi-line Treatment (Including Immunotherapy)
Brief Title: The Efficacy and Safety of Sintilimab in Combination With Multimodal Radiotherapy in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Collaborators: Chengdu City No.2 People's Hospital (Unknown); No.3 People's Hospital of Chengdu (Unknown); Sichuan Provincial People's Hospital (Other); The First People's Hospital of Ziyang (Unknown); No.5 People's Hospital of Chengdu (Unknown)
Responsible Party: Principal Investigator, Xingchen Peng, Associate Professor and Doctoral Advisor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX20210601
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Sintilimab; nasopharyngeal carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — sintilimab

STUDY DESIGN:
Intervention Model Description: Sintilimab in combination with Multimodality Radiotherapy group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab in combination with Multimodality Radiotherapy group (Experimental): The dose of sintilimab was 200mg per dose, intravenously, once every 3 weeks. Multimodal radiotherapy methods: ①SBRT: ≥1 independent lesion was selected, with a single dose of 8-10Gy and a total dose of 40-60Gy, divided into 5-6 times of radiotherapy. The final frequency and total dose of radiotherapy were determined by the radiologist.② Low-dose radiotherapy: ≥1 independent lesion was selected, and the single dose, the final frequency of radiotherapy and the total dose were determined by the radiologist.
  Interventions: Drug: Sintilimab in combination with Multimodality Radiotherapy

INTERVENTIONS:
Drug: Sintilimab in combination with Multimodality Radiotherapy — Participants will be treated with sintilimab in combination with multimodality radiotherapy

SUMMARY:
Nasopharyngeal carcinoma is the most common malignant tumor of head and neck in southern China. After standard treatment, about 20% of the patients had local recurrence or distant metastasis, and the patients faced death in a short time. Currently, there is no recommended treatment for patients with recurrent or metastatic nasopharyngeal carcinoma who have unsatisfactory results of first-line chemotherapy and subsequent immunotherapy. Patients who have failed multiline therapy have a low survival rate and no drugs are available.This project aims to evaluate the efficacy and safety of sintilimab in combination with multimodal radiotherapy for patients with recurrent or metastatic nasopharyngeal carcinoma who have previously received immunotherapy and still progress after multiline therapy, and to seek a new therapeutic approach for such patients.

ELIGIBILITY:
Inclusion Criteria:

1. The histopathological diagnosis was recurrent or distant metastatic nasopharyngeal carcinoma;
2. Have received two or more lines of treatment, including at least one immunocheckpoint inhibitor related therapy containing PD-1/L1, and have achieved clinical benefit;
3. Aged between 18 and 65 at the date of signing the informed consent;
4. ECOG score 0-1;
5. At least ≥1 measurable lesion according to Recist v1.1, or ≥1 measurable lesion with definite progression after local treatment (based on Recist v1.1 criteria);At the same time, there were more than 1 radiotherapy foci and lesions with radiographic evaluation of distant effect.
6. Life expectancy ≥12 weeks;
7. Major organ functions within 28 days prior to treatment meet the following criteria:

A. Routine blood test criteria (without blood transfusion within 14 days) : hemoglobin (Hb) ≥80g/L;Neutrophils absolute value (ANC) ≥1.5×109/L;Platelet (PLT) ≥80×109/L; B. Biochemical tests should meet the following criteria: total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN);Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN, if accompanied by liver metastasis, ALT and AST≤5×ULN;Serum creatinine (CR) ≤1.5×ULN or creatinine clearance rate (CCR)≥60ml/min; C. Coagulograms should meet the following criteria: International Standardized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5ULN;Activated partial thromboplastin time (APTT) ≤1.5 ULN (if the patient is receiving anticoagulant therapy, as long as PT and APTT are within the expected treatment range); D. centrifuge markers and urinary natriuretic peptide (BNP) ≤ULN; E. Thyroid function: T3 and T4 levels were normal after medication; 8. Women of reproductive age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and for 120 days after the end of the study;Negative serum or urinary pregnancy test within 7 days prior to study enrollment; 9. With my consent and signed the informed consent.

Exclusion Criteria:

1. Previous use of immunocheckpoint inhibitors combined with radiotherapy after recurrence and metastasis;
2. A history of other malignant tumors within the previous 5 years or at the same time, except cured basal cell carcinoma of the skin, carcinoma in situ of the cervix and papillary carcinoma of the thyroid;
3. known allergic reactions to active ingredients of PD-1 monoclonal antibody or any excipients;
4. Symptomatic central nervous system metastasis;
5. Those who had received potent CYP3A4 inhibitor treatment within one week before enrollment, or inducer CYP3A4 treatment within two weeks before enrollment;
6. The New York Heart Association's cardiac function classification is Grade III-IV congestive heart failure;
7. An ischemic cardiovascular event occurred within 1 year prior to treatment;
8. QT interval of ECG >500 ms;
9. Have received systemic immunosuppressive therapy;
10. Participate in clinical trials of other interventional drugs within 4 weeks before the first administration;
11. Subjects who require systematic treatment with corticosteroids (greater than 10mg equivalent daily dose of prednisone) or other immunosuppressant within 2 weeks prior to the first use of the study drug;
12. Have received an anti-tumor vaccine or a live vaccine within 4 weeks before the first administration of the investigational drug;
13. Major surgery or severe trauma within 4 weeks before the first use of the study drug;
14. Severe infections (CTCAE > grade 2) occurred within 4 weeks before the first use of the study drug, such as severe pneumonia, bacteremia, infection complications, etc., requiring hospitalization;Baseline chest imaging examination suggests active pulmonary inflammation, signs and symptoms of infection within 2 weeks prior to the first use of the study drug, or the need for oral or intravenous antibiotic treatment (excluding prophylactic use of antibiotics);
15. Have a history of active autoimmune diseases or autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, pituitaritis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases and syndromes);Autoimmune-mediated hypothyroidism treated with a steady dose of thyroid-replacement hormone and with a steady dose of insulin in type 1 diabetes were included;This does not include patients with vitiligo or cured childhood asthma/allergies who do not need any intervention as adults;
16. Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation or bone marrow transplantation;
17. History of non-infectious pneumonia
18. Patients with active tuberculosis infection found by medical history or CT examination, or patients with active tuberculosis infection found within 1 year before enrollment, or patients with active tuberculosis infection found before 1 year but without formal treatment;
19. Subsubjects had active hepatitis (HBV DNA≥2000IU/ mL or 10000 copies/ mL) and hepatitis C (HCV antibody positive and HCV-RNA above the detection limit of the assay method);
20. A history of known abuse of psychotropic substances, alcoholism and drug abuse;
21. Being pregnant or lactating;
22. There is any history, disease, treatment, or abnormal laboratory result that may interfere with the results of the study and prevent subjects from participating fully in the study, or the investigator deems that participation is not in the best interest of the subjects.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | up to approximately 2 years

SECONDARY OUTCOMES:
Progression-free survival | up to approximately 2 years
Overall survival | up to approximately 2 years
Duration of remission | up to approximately 2 years
1 year overall survival | 1 years after treatment finished
Adverse reactions | Time Frame: from the first drug administration to within 30 days for the last therapy

IPD SHARING:
Plan to Share IPD: No